CLINICAL TRIAL: NCT01871350
Title: Effects of Chemotherapy and Nutritional Intervention on Gut Function and Metabolism in Cancer
Brief Title: Nutrition Intervention During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-0504
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cancer Patients Receiving Chemotherapy or Chemoradiotherapy
Keywords: Cancer; Chemotherapy; Chemo related toxicity; Protein digestion; Fat digestion; Gut function; Glucose absorption; Muscle function
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein and Fish Oil (Experimental): Low Dose (FFM <49kg): 30.00g milk protein + 12.75g maltodextrin and 6g fish oil
  High dose (FFM >49kg): 40.00g milk protein + 17.00g maltodextrin and 8g fish oil
  Interventions: Dietary Supplement: Daily intake for 10 weeks (+/- 2 weeks)
- Protein (Experimental): Low Dose (FFM <49kg): 30.00g milk protein + 12.75g maltodextrin and 6g olive oil
  High dose (FFM >49kg): 40.00g milk protein + 17.00g maltodextrin and 8g olive oil
  Interventions: Dietary Supplement: Daily intake for 10 weeks (+/- 2 weeks)
- Placebo (Placebo Comparator): Low Dose (FFM <49kg): 12.75g maltodextrin and 6g olive oil
  High dose (FFM >49kg): 17.00g maltodextrin and 8g olive oil
  Interventions: Dietary Supplement: Daily intake for 10 weeks (+/- 2 weeks)

INTERVENTIONS:
Dietary Supplement: Daily intake for 10 weeks (+/- 2 weeks)

SUMMARY:
Weight loss and muscle wasting commonly occurs in patients with cancer, negatively influencing their quality of life, treatment response and survival. Weight loss has been reported as a side effect of chemotherapy treatment in cancer. Weight changes may be the consequence of energy imbalance and disturbances in protein metabolism (through different factors linked with chemotherapy), such as reduced caloric and protein intake (partly related to depression), poor treatment tolerance, hormonal alterations, systemic inflammation etc. This results in body composition modiﬁcations in favor of fat gain and/or lean body mass loss in early stage cancer and loss of both fat mass and lean mass in advanced cancer. Depletion of lean tissue in cancer patients is related to short survival, and decreased skeletal muscle mass and function may result in fatigue and inactivity, which contributes to fat mass changes and can be responsible for chemo-toxicity and increased mortality.

Gains in muscle mass are difficult to achieve in cancer unless specific metabolic abnormalities are targeted. Recently, the investigators observed that essential amino acid mixtures (EAA) are able to induce protein anabolism in patients with stage III and IV non-small cell lung cancer. Previous experimental research and clinical studies in cachectic conditions (including cancer) indicate that polyunsaturated fatty acids (PUFA) are able to attenuate protein degradation by improving the anabolic response to feeding and by decreasing the acute phase response. Eicosapentaenoic acid (EPA) (in combination with docosahexaenoic acid (DHA)) has been shown to effectively inhibit weight loss in several disease states; however, weight and muscle mass gain was not present or minimal. Recent studies examining the effect of fish oil supplementation in relation to chemotherapy have been inconclusive but found potential beneficial effects on physical performance and increased efficacy of first-line chemotherapy in patients with non-small cell lung cancer.

It is the investigators' hypothesis that supplementation with milk protein (containing essential amino acids) carbohydrate (CHO) mixture in combination with fish oil supplementation will target the metabolic alterations in cancer patients receiving chemotherapy, attenuating the negative effects of chemotherapy on gut function, muscle mass and muscle function, and cognition; and leading to reduced toxicity from chemotherapy.

DETAILED DESCRIPTION:
For the cancer subjects, the study involves 1 test day prior to a chemotherapy treatment, a 10-week (± 2 weeks) nutritional intervention period at home starting the first day of the chemotherapy treatment, and one test day after this intervention. Chemotherapy in general lasts at least a few months. Recent studies indicate that a 10-week nutritional supplementation period should be long enough to reach significant improvements in nutritional and clinical outcome parameters during chemotherapy. Throughout these 10 weeks the cancer subjects will take the supplements at home. Cancer subjects will be randomly assigned to receive either fish oil or a placebo and protein or a placebo and will take these supplements daily throughout 10 weeks during chemotherapy.

For the healthy subjects, the study will involve one test day (approx. 8 hours).

On the test days, the response to a protein meal will be examined and subjects will receive a mixture of amino acids which are a little bit heavier than normal, called stable isotopes. Subjects will also ingest a sugar drink to assess gut permeability. In total, approximate 120 ml of blood will be drawn on each test day to assess outcome measures. The investigators' will also collect urine over these 8 hours, and cancer subjects are asked to collect a fecal sample the day before the test day.

After completing the nutritional intervention study, cancer subjects will be monitored for up to 6 months via 2 phone calls and through their physician as part of clinical care. Between 6 months and 2 years after completion of the study, information about disease progression (survival) will be obtained from the physician.

ELIGIBILITY:
Inclusion criteria cancer subjects:

* Diagnosed with cancer
* Scheduled for chemotherapy or chemoradiotherapy
* Ability to sign informed consent
* Age 18y and older
* Ability to lie in supine position for 7 hours

Inclusion criteria healthy subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Age 18 years or older
* No diagnosis of cancer

Exclusion Criteria

* Presence of fever within the last 3 days
* BMI > 38 kg/m2 (healthy controls only)
* Untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Use of protein or amino acid containing nutritional supplements within 5 days of first test day
* Known hypersensitivity to fish and/or shellfish, Swanson EFAs Super EPA Fish oil or any of its ingredients, Swanson EFAs Certified Organic Extra Virgin Olive oil or any of its ingredients, Smartfish Nutrifriend or any of its ingredients (Cancer subjects only)
* Use of supplements containing EPA+DHA 3 months prior to the first test day
* Any other condition according to the PI or nurse that would interfere with the study or safety of the patient
* Failure to give informed consent
* (Possible) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2015-11-03 (Actual); Study Completion 2015-11-03 (Actual)

PRIMARY OUTCOMES:
Net whole-body protein synthesis | Acutely before and after 4 hours of feeding and the change after 10 weeks of supplementation
  The acute change in whole-body protein synthesis rate before and after intake of meal is determined on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.

SECONDARY OUTCOMES:
Citrulline Rate of appearance | In the postabsorptive state for 4h on the first test day and the change on the second test day after 10 weeks of supplementation
  Plasma enrichment of citrulline is determined on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Glucose absorption | 7 hours during the test day and the change after 10 weeks of supplementation
  Recovery of 3-O-Methyl-D-glucose in the urine is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Gut permeability | 7 hours during the test day and the change after 10 weeks of supplementation
  Recovery of rhamnose/lactulose in urine is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Skeletal and respiratory muscle strength | In the postabsorptive state on the first test day and the change on the second test day after 10 weeks of supplementation
  Difference in leg strength and fatigue, handgrip strength and fatigue, and inspiratory and expiratory pressure between heart failure patients and healthy controls on test day 1. The cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Cognitive function | On the first test day and the change on the second test day after 10 weeks of supplementation
  Outcome of neuro-psychological tests in heart failure patients and healthy controls in relation to the tryptophan metabolism. The cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Fatty acid digestion after feeding | Acutely after 4 hours of feeding and the change after 10 weeks of supplementation
  Enrichment in palmitic acid and tripalmitin fatty acids in plasma in response to a meal is measured on the first test day in for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Protein digestion after feeding | Acutely after 4 hours of feeding and the change after 10 weeks of supplementation
  Ratio enrichment free phenylalanine vs phenylalanine from protein spirulina in response to a meal is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Whole body collagen breakdown rate | In the postabsorptive state on the first test day and the change on the second test day after 10 weeks of supplementation
  Hydroxyproline enrichment in plasma is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Tryptophan turnover rate | In the postabsorptive state on the first test day and the change on the second test day after 10 weeks of supplementation
  Tryptophan enrichment in plasma is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Insulin response to feeding | Before and acutely after 4 hours of feeding and the change after 10 weeks of supplementation
  The acute change in insulin levels before and after intake of meal is determined on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Fat-free mass | In postabsorptive state on test day 1 and the difference on test day 2, after 10 weeks of supplementation
  Fat free mass is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Myofibrillar protein breakdown rate | Before and acutely after 4 hours of feeding and the change after 10 weeks of supplementation
  The acute change 3-methylhistidine enrichment in plasma before and after intake of meal is determined on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Glycine rate of appearance | In the postabsorptive state on the first test day and the change on the second test day after 10 weeks of supplementation
  Glycine enrichment in plasma is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Taurine turnover rate | In the postabsorptive state on the first test day and the change on the second test day after 10 weeks of supplementation
  Enrichment of taurine in plasma is measured on the first test day for the healthy control group and the cancer group. Secondly, the cancer patients in all 3 intervention arms are also measured after 10 weeks of intervention to examine the effects of fish oil and protein supplementation during chemotherapy on this outcome measure.
Functional Status | On the first test day and the change on the second test day after 10 weeks of supplementation
  Functional status will be assessed by the Karnofsky Performance Score, a widely used method to assess the functional status of a cancer patient. It describes a patient's functional status as a comprehensive 11-point scale ranging from 0% to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle PKJ Engelen, PhD, Principal Investigator — Texas A&M Univeristy
Locations (1):
- Texas A&M University, College Station, Texas, United States